CLINICAL TRIAL: NCT01097655
Title: Use of KALETRA® Tablets in Adult HIV-infected Patients: Data From the Multicenter Star/Stella Cohort
Brief Title: Study on the Usage, Dosing, Tolerability, and Effectiveness of Kaletra Tablet
Status: Completed | Type: Observational
Sponsor: AbbVie (prior sponsor, Abbott) (Industry)
Collaborators: Veeda Clinical Research (Industry)
Responsible Party: Sponsor
Organization: AbbVie (Industry)
Other Study IDs: P06-131
Record Dates: First submitted 2010-02-26; First posted 2010-04-02 (Estimated); Results first posted 2017-05-23 (Actual); Last update posted 2017-05-23 (Actual); Status verified 2017-05

CONDITIONS: Human Immunodeficiency Virus
Keywords: Tablets; Infection; Non Nucleoside Reverse Transcriptase Inhibitor; Tolerability; Viral load; Human immunodeficiency Virus; Effectiveness; Treatment-naïve
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- HIV-infected Participants: HIV-infected participants starting with Kaletra tablets.
  Participants included 3 subgroups:
  * antiretroviral therapy (ART) treatment-naïve participants starting with Kaletra tablets
  * participants receiving their first protease inhibitor (PI)-containing regimen (apart from Kaletra) pretreated with any non nucleoside reverse transcriptase inhibitor (NNRTI)-containing or nucleoside reverse transcriptase inhibitor (NRTI)-containing regimen
  * participants pretreated with a PI-containing regimen (apart from Kaletra).

SUMMARY:
The objective of this study is to observe and collect data on the usage, dosing, tolerability, and effectiveness of Kaletra (lopinavir/ritonavir) tablets in human immunodeficiency virus (HIV)-infected patients. In some patients, the study is to show the impact on tolerability of changing therapy to Kaletra tablets from other regimens.

DETAILED DESCRIPTION:
This study was designed as a non-interventional observational study. Kaletra was prescribed in the usual manner in accordance with the terms of the local market authorization with regards to dose, population and indication as well as local guidelines.

ELIGIBILITY:
Inclusion Criteria:

* Patients with HIV infection
* Patients that will be treated with Kaletra tablets independent from their participation in this study

Exclusion Criteria:

* Hypersensitivity against Kaletra or other ingredients
* Severe liver insufficiency
* No concommitant astemizole, terfenadine, oral midazolam, triazolam, cisapride, pimozide, amiodarone, ergotamine, dihydroergotamine, ergometrine, methylergometrine, vardenafil and St. John's wort
* Patients who received more than 1 protease inhibitor during their therapy history

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: * Community sample; HIV-infected patients
  * For Belgium: AIDS references centers (probability sample)
Sampling Method: Non-Probability Sample
Enrollment: 3049 (Actual)
Dates: Start 2006-08; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sandra Bloch, MD, Study Director — AbbVie Deutschland GmbH & Co. KG, Medical Department

REFERENCES:
- See also: Related Info — http://rxabbvie.com

RESULTS

PARTICIPANT FLOW:
Groups:
- HIV-infected Participants: HIV-infected participants starting with Kaletra tablets.
Period: Overall Study
Arm/Group | HIV-infected Participants
Started | 3049
Completed | 3039 (participants included for analysis)
Not Completed | 10
Not completed — Withdrawal by Subject | 1
Not completed — Subject Documented Twice | 1
Not completed — Did Not Meet Inclusion Criteria | 8

BASELINE CHARACTERISTICS:
Arm/Group | HIV-infected Participants
Number analyzed (Participants) | 3039
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: participants with age recorded at Baseline
  years
    number analyzed (Participants) | 2896
    (all) | 40.7 (10.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 595
  Male | 2444

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Absolute Cluster of Differentiation 4 (CD4) Cell Count
Description: Changes in participants' CD4 cell counts were assessed by measuring the change from Baseline in the number of CD4 cells at scheduled visits planned as part of routine care.
Time Frame: Baseline (Week 0) to Week 144
Population: Participants with an assessment at Baseline. Number analyzed=participants with an assessment at given time point.
Measure: Mean (Standard Deviation); unit: cells/μL
Arm/Group | HIV-infected Participants
Number analyzed (Participants) | 2981
cells/μL
  Change at Week 4: number analyzed (Participants) | 2378
  Change at Week 4 | 99.8 (145.2)
  Change at Week 12: number analyzed (Participants) | 2391
  Change at Week 12 | 133.3 (148.7)
  Change at Week 24: number analyzed (Participants) | 2240
  Change at Week 24 | 160.5 (177.6)
  Change at Week 36: number analyzed (Participants) | 2004
  Change at Week 36 | 185.9 (181.2)
  Change at Week 48: number analyzed (Participants) | 1867
  Change at Week 48 | 213.6 (225.1)
  Change at Week 60: number analyzed (Participants) | 1694
  Change at Week 60 | 228.4 (204.6)
  Change at Week 72: number analyzed (Participants) | 1545
  Change at Week 72 | 250.1 (205.1)
  Change at Week 84: number analyzed (Participants) | 1370
  Change at Week 84 | 263.8 (214.8)
  Change at Week 96: number analyzed (Participants) | 1340
  Change at Week 96 | 276.3 (212.8)
  Change at Week 108: number analyzed (Participants) | 1222
  Change at Week 108 | 291.0 (247.6)
  Change at Week 120: number analyzed (Participants) | 1171
  Change at Week 120 | 294.3 (216.5)
  Change at Week 132: number analyzed (Participants) | 1110
  Change at Week 132 | 303.8 (229.3)
  Change at Week 144: number analyzed (Participants) | 1173
  Change at Week 144 | 316.1 (228.2)

2. Primary Outcome: Change From Baseline in HIV-1 Ribonucleic Acid (RNA) Viral Load
Description: Changes in participants' HIV-1 RNA viral load were assessed by measuring the change from Baseline at scheduled visits planned as part of routine care.
Time Frame: Baseline (Week 0) to Week 144
Population: Participants with an assessment at Baseline. Number analyzed=participants with an assessment at given time point.
Measure: Mean (Standard Deviation); unit: log copies/mL
Arm/Group | HIV-infected Participants
Number analyzed (Participants) | 2959
log copies/mL
  Change at Week 4: number analyzed (Participants) | 2323
  Change at Week 4 | -1.90 (0.97)
  Change at Week 12: number analyzed (Participants) | 2296
  Change at Week 12 | -2.53 (1.23)
  Change at Week 24: number analyzed (Participants) | 2089
  Change at Week 24 | -2.83 (1.35)
  Change at Week 36: number analyzed (Participants) | 1821
  Change at Week 36 | -2.89 (1.40)
  Change at Week 48: number analyzed (Participants) | 1693
  Change at Week 48 | -2.89 (1.41)
  Change at Week 60: number analyzed (Participants) | 1532
  Change at Week 60 | -2.93 (1.38)
  Change at Week 72: number analyzed (Participants) | 1377
  Change at Week 72 | -2.92 (1.36)
  Change at Week 84: number analyzed (Participants) | 1230
  Change at Week 84 | -2.92 (1.37)
  Change at Week 96: number analyzed (Participants) | 1198
  Change at Week 96 | -2.93 (1.38)
  Change at Week 108: number analyzed (Participants) | 1093
  Change at Week 108 | -2.93 (1.39)
  Change at Week 120: number analyzed (Participants) | 1070
  Change at Week 120 | -2.92 (1.36)
  Change at Week 132: number analyzed (Participants) | 999
  Change at Week 132 | -2.94 (1.36)
  Change at Week 144: number analyzed (Participants) | 1049
  Change at Week 144 | -2.97 (1.34)

3. Other Pre Specified Outcome: Prevalence of Adverse Events (Weeks 0-144), Per Event
Description: Percentage of overall number of adverse events experienced during Weeks 0-144 by adverse event type. Doctors asked participants for adverse events, grouped them into categories given in the electronic case report form (eCRF). The list of adverse events included in the eCRF were hypertriglyceridemia, hypercholesterolemia, low high density lipoprotein (HDL) cholesterol, high low density lipoprotein (LDL) cholesterol, hyperglycemia, hyperbilirubinemia, elevated aspartate aminotransferase (AST), elevated alanine aminotransferase (ALT), elevated gamma glutamyl transferase (γGT), elevated alkaline phosphatase, stomatitis, nausea, vomiting, diarrhea, abdominal pain, mood disorder, neurocerebellar disorder, neurocontrol disorder, headache, fatigue, fever, other (listed as 'not specified').
Time Frame: Weeks 0 to 144
Measure: Number; unit: percentage of adverse events
Units Other Than Participants: Adverse Events
Arm/Group | HIV-infected Participants
Number analyzed (Participants) | 3039
Number analyzed (Adverse Events) | 44499
percentage of adverse events
  Hypertriglyceridemia | 12.4
  Hypercholesterolemia | 19.3
  Low HDL Cholesterol | 0.5
  High LDL Cholesterol | 2.3
  Hyperglycemia | 3.0
  Hyperbilirubinemia | 2.7
  Elevated AST | 3.5
  Elevated ALT | 4.1
  Elevated γGT | 7.3
  Elevated Alkaline Phosphatase | 3.1
  Stomatitis | 0.6
  Nausea | 4.2
  Vomiting | 1.5
  Diarrhea | 18.3
  Abdominal Pain | 2.9
  Mood Disorder | 5.0
  Neurocerebellar Disorder | 0.6
  Neurocontrol Disorder | 0.0
  Headache | 1.9
  Fatigue | 4.0
  Fever | 1.4
  Not Specified | 4.8

4. Other Pre Specified Outcome: Prevalence of Adverse Events (Weeks 0-144), Per Participant
Description: Percentage of participants who experienced at least 1 adverse event during Weeks 0-144 by adverse event type. Doctors asked participants for adverse events, grouped them into categories given in the eCRF. The list of adverse events included in the eCRF were hypertriglyceridemia, hypercholesterolemia, low HDL cholesterol, high LDL cholesterol, hyperglycemia, hyperbilirubinemia, elevated AST, elevated ALT, elevated γGT, elevated alkaline phosphatase, stomatitis, nausea, vomiting, diarrhea, abdominal pain, mood disorder, neurocerebellar disorder, neurocontrol disorder, headache, fatigue, fever, other (listed as 'not specified').
Time Frame: Weeks 0 to 144
Measure: Number; unit: percentage of participants
Arm/Group | HIV-infected Participants
Number analyzed (Participants) | 3039
percentage of participants
  Hypertriglyceridemia | 14.1
  Hypercholesterolemia | 16.3
  Low HDL Cholesterol | 1.6
  High LDL Cholesterol | 4.0
  Hyperglycemia | 5.8
  Hyperbilirubinemia | 3.9
  Elevated AST | 6.7
  Elevated ALT | 7.5
  Elevated γGT | 9.3
  Elevated Alkaline Phosphatase | 4.7
  Stomatitis | 2.0
  Nausea | 11.5
  Vomiting | 4.6
  Diarrhea | 32.7
  Abdominal Pain | 8.0
  Mood Disorder | 9.0
  Neurocerebellar Disorder | 1.7
  Neurocontrol Disorder | 0.0
  Headache | 5.2
  Fatigue | 8.7
  Fever | 4.4
  Not Specified | 30.4

ADVERSE EVENTS:
Time Frame: Through Week 144
Description: Serious adverse events only were collected and coded by MedDRA. Per protocol, the number of participants with events were collected for each event, but from the source documentation to tell how many of the participants are counted in more than one adverse event (i.e., it is not possible to compute the Total Number of Participants Affected). Please see Outcome Measures 3 and 4 for these data.
Arm/Group | HIV-infected Participants
Serious Adverse Events (participants affected / at risk) | 79/3039
Other Adverse Events (participants affected / at risk) | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | HIV-infected Participants (N=3039)
ANAEMIA (Blood and lymphatic system disorders) | 3
EOSINOPHILIA (Blood and lymphatic system disorders) | 1
HAEMOLYTIC ANAEMIA (Blood and lymphatic system disorders) | 1
LYMPHADENITIS (Blood and lymphatic system disorders) | 1
LYMPHADENOPATHY (Blood and lymphatic system disorders) | 1
MACROCYTOSIS (Blood and lymphatic system disorders) | 1
PANCYTOPENIA (Blood and lymphatic system disorders) | 2
PLASMACYTOSIS (Blood and lymphatic system disorders) | 1
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 1
ANGINA PECTORIS (Cardiac disorders) | 1
ARTERIOSCLEROSIS CORONARY ARTERY (Cardiac disorders) | 1
ATRIOVENTRICULAR BLOCK (Cardiac disorders) | 1
ATRIOVENTRICULAR BLOCK SECOND DEGREE (Cardiac disorders) | 1
ATRIOVENTRICULAR DISSOCIATION (Cardiac disorders) | 1
BRADYCARDIA (Cardiac disorders) | 1
BUNDLE BRANCH BLOCK RIGHT (Cardiac disorders) | 1
CARDIAC VALVE DISEASE (Cardiac disorders) | 1
DEGENERATIVE MITRAL VALVE DISEASE (Cardiac disorders) | 1
EXTRASYSTOLES (Cardiac disorders) | 1
MYOCARDIAL INFARCTION (Cardiac disorders) | 2
PLEUROPERICARDITIS (Cardiac disorders) | 1
RIGHT VENTRICULAR FAILURE (Cardiac disorders) | 1
VENTRICULAR TACHYCARDIA (Cardiac disorders) | 1
HYPERTHYROIDISM (Endocrine disorders) | 1
EYE SWELLING (Eye disorders) | 1
ABDOMINAL HERNIA (Gastrointestinal disorders) | 1
ABDOMINAL PAIN (Gastrointestinal disorders) | 5
ALCOHOLIC PANCREATITIS (Gastrointestinal disorders) | 1
ANAL FISTULA (Gastrointestinal disorders) | 2
ASCITES (Gastrointestinal disorders) | 1
CHRONIC GASTRITIS (Gastrointestinal disorders) | 1
DIARRHOEA (Gastrointestinal disorders) | 6
DIARRHOEA HAEMORRHAGIC (Gastrointestinal disorders) | 1
DYSPHAGIA (Gastrointestinal disorders) | 1
GASTROINTESTINAL DISORDER (Gastrointestinal disorders) | 1
GINGIVITIS ULCERATIVE (Gastrointestinal disorders) | 1
HAEMATEMESIS (Gastrointestinal disorders) | 1
HAEMORRHOIDS (Gastrointestinal disorders) | 2
INGUINAL HERNIA (Gastrointestinal disorders) | 2
LEUKOPLAKIA ORAL (Gastrointestinal disorders) | 1
NAUSEA (Gastrointestinal disorders) | 4
OESOPHAGITIS (Gastrointestinal disorders) | 1
PANCREATIC CYST (Gastrointestinal disorders) | 1
PANCREATITIS (Gastrointestinal disorders) | 1
PROCTALGIA (Gastrointestinal disorders) | 1
SALIVARY GLAND CYST (Gastrointestinal disorders) | 1
VOMITING (Gastrointestinal disorders) | 3
ASTHENIA (General disorders) | 1
CHEST PAIN (General disorders) | 1
CHILLS (General disorders) | 1
DRUG INTOLERANCE (General disorders) | 1
DRUG WITHDRAWAL SYNDROME (General disorders) | 1
GENERAL PHYSICAL HEALTH DETERIORATION (General disorders) | 4
PAIN (General disorders) | 3
PYREXIA (General disorders) | 5
HEPATIC CIRRHOSIS (Hepatobiliary disorders) | 1
HEPATIC LESION (Hepatobiliary disorders) | 1
IMMUNE RECONSTITUTION INFLAMMATORY SYNDROME (Immune system disorders) | 2
AIDS DEMENTIA COMPLEX (Infections and infestations) | 1
ACQUIRED IMMUNODEFICIENCY SYNDROME (Infections and infestations) | 1
ANAL ABSCESS (Infections and infestations) | 1
CHLAMYDIAL INFECTION (Infections and infestations) | 1
CYTOMEGALOVIRUS COLITIS (Infections and infestations) | 1
ENDOCARDITIS (Infections and infestations) | 1
FUNGAL OESOPHAGITIS (Infections and infestations) | 1
GASTROENTERITIS (Infections and infestations) | 2
GASTROINTESTINAL INFECTION (Infections and infestations) | 2
HELICOBACTER GASTRITIS (Infections and infestations) | 1
HERPES VIRUS INFECTION (Infections and infestations) | 1
HERPES ZOSTER (Infections and infestations) | 2
LEISHMANIASIS (Infections and infestations) | 1
LYMPH NODE TUBERCULOSIS (Infections and infestations) | 1
LYMPHOGRANULOMA VENEREUM (Infections and infestations) | 1
MYCOBACTERIUM AVIUM COMPLEX INFECTION (Infections and infestations) | 1
OESOPHAGEAL CANDIDIASIS (Infections and infestations) | 1
OPHTHALMIC HERPES ZOSTER (Infections and infestations) | 1
ORAL CANDIDIASIS (Infections and infestations) | 1
ORAL HERPES (Infections and infestations) | 1
PNEUMOCYSTIS JIROVECII PNEUMONIA (Infections and infestations) | 1
PNEUMONIA (Infections and infestations) | 5
PULMONARY TUBERCULOSIS (Infections and infestations) | 2
SALMONELLOSIS (Infections and infestations) | 1
SECONDARY TRANSMISSION (Infections and infestations) | 1
SINUSITIS (Infections and infestations) | 1
STAPHYLOCOCCAL SEPSIS (Infections and infestations) | 1
TONSILLITIS (Infections and infestations) | 1
FALL (Injury, poisoning and procedural complications) | 1
FEMORAL NECK FRACTURE (Injury, poisoning and procedural complications) | 1
LUMBAR VERTEBRAL FRACTURE (Injury, poisoning and procedural complications) | 3
BLOOD TRIGLYCERIDES INCREASED (Investigations) | 2
CYTOMEGALOVIRUS TEST POSITIVE (Investigations) | 1
GENERAL PHYSICAL CONDITION ABNORMAL (Investigations) | 1
WEIGHT DECREASED (Investigations) | 1
DECREASED APPETITE (Metabolism and nutrition disorders) | 1
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 1
INGUINAL MASS (Musculoskeletal and connective tissue disorders) | 1
INTERVERTEBRAL DISC PROTRUSION (Musculoskeletal and connective tissue disorders) | 3
OSTEONECROSIS (Musculoskeletal and connective tissue disorders) | 1
OSTEOPOROSIS (Musculoskeletal and connective tissue disorders) | 1
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 1
SPINAL PAIN (Musculoskeletal and connective tissue disorders) | 1
ANAL CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
ANAPLASTIC LARGE CELL LYMPHOMA T- AND NULL-CELL TYPE STAGE IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
ANOGENITAL WARTS (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
BURKITT'S LYMPHOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3
EXTRANODAL MARGINAL ZONE B-CELL LYMPHOMA (MALT TYPE) (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
HEPATIC CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
KAPOSI'S SARCOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
PAPILLOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
PLASMABLASTIC LYMPHOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
ATAXIA (Nervous system disorders) | 1
BALANCE DISORDER (Nervous system disorders) | 1
CEREBRAL ARTERIOSCLEROSIS (Nervous system disorders) | 1
CEREBRAL ATROPHY (Nervous system disorders) | 1
CEREBRAL INFARCTION (Nervous system disorders) | 2
DISTURBANCE IN ATTENTION (Nervous system disorders) | 1
FACIAL PARESIS (Nervous system disorders) | 1
HEADACHE (Nervous system disorders) | 3
HYPOAESTHESIA (Nervous system disorders) | 1
MEMORY IMPAIRMENT (Nervous system disorders) | 1
MENINGEAL DISORDER (Nervous system disorders) | 1
PARAESTHESIA (Nervous system disorders) | 1
RADICULOPATHY (Nervous system disorders) | 1
SOMNOLENCE (Nervous system disorders) | 1
ABORTION (Pregnancy, puerperium and perinatal conditions) | 1
ABORTION MISSED (Pregnancy, puerperium and perinatal conditions) | 1
ABORTION SPONTANEOUS (Pregnancy, puerperium and perinatal conditions) | 3
MATERNAL CONDITION AFFECTING FOETUS (Pregnancy, puerperium and perinatal conditions) | 1
PLACENTAL INSUFFICIENCY (Pregnancy, puerperium and perinatal conditions) | 1
PREMATURE BABY (Pregnancy, puerperium and perinatal conditions) | 1
APATHY (Psychiatric disorders) | 1
CONFUSIONAL STATE (Psychiatric disorders) | 1
DELIRIUM (Psychiatric disorders) | 1
DEPRESSION (Psychiatric disorders) | 1
DISORIENTATION (Psychiatric disorders) | 1
HYDRONEPHROSIS (Renal and urinary disorders) | 1
NEPHROLITHIASIS (Renal and urinary disorders) | 1
NOCTURIA (Renal and urinary disorders) | 1
RENAL CYST (Renal and urinary disorders) | 1
RENAL FAILURE (Renal and urinary disorders) | 1
URINARY BLADDER POLYP (Renal and urinary disorders) | 1
ADENOMYOSIS (Reproductive system and breast disorders) | 1
MENOMETRORRHAGIA (Reproductive system and breast disorders) | 1
PROSTATIC MASS (Reproductive system and breast disorders) | 1
VAGINAL HAEMORRHAGE (Reproductive system and breast disorders) | 2
CHRONIC OBSTRUCTIVE PULMONARY DISEASE (Respiratory, thoracic and mediastinal disorders) | 1
COUGH (Respiratory, thoracic and mediastinal disorders) | 1
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 3
LUNG INFILTRATION (Respiratory, thoracic and mediastinal disorders) | 1
OROPHARYNGEAL PAIN (Respiratory, thoracic and mediastinal disorders) | 1
RALES (Respiratory, thoracic and mediastinal disorders) | 1
ABORTION INDUCED (Surgical and medical procedures) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
AbbVie requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. AbbVie requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if AbbVie needs to secure patent or proprietary protection.